CLINICAL TRIAL: NCT03101085
Title: S-Equol in Alzheimer's Disease 2 (SEAD2) Trial
Brief Title: S-Equol in Alzheimer's Disease 2 Trial
Acronym: SEAD2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Russell Swerdlow (Other)
Collaborators: Ausio Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor-Investigator, Russell Swerdlow, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SEAD2; SEAD2 (Other Grant/Funding Number: Ausio (Solely funded by Ausio; was not an NIH-funded study))
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Equol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- S-equol First, Then Placebo (Other): In this arm, participants receive S-equol 50mg twice daily for one month, followed by placebo twice daily for one month. There was no washout period.
  Interventions: Drug: S-equol and Placebo
- Placebo First, Then S-equol (Other): In this arm, participants receive placebo twice daily for one month, followed by S-equol 50mg twice daily for one month. There was no washout period.
  Interventions: Drug: Placebo and S-equol

INTERVENTIONS:
Drug: S-equol and Placebo — S-equol is an estrogen receptor β (ERβ) agonist. Provided in capsules. The placebo is a matched pill that cannot be distinguished from the active S-equol.
  Other Names: S-equol is also called AUS-131
  Arms: S-equol First, Then Placebo
Drug: Placebo and S-equol — S-equol is an estrogen receptor β (ERβ) agonist. Provided in capsules. The placebo is a matched pill that cannot be distinguished from the active S-equol.
  Other Names: S-equol is also called AUS-131
  Arms: Placebo First, Then S-equol

SUMMARY:
By doing this study researchers hope to learn if S-equol, a compound that acts like estrogen in the body, causes an increase in mitochondrial activity. Researchers also hope to determine the safety and tolerability of a therapeutic dose of S-equol and whether or not it influences cognition.

DETAILED DESCRIPTION:
Enrolled participants with a diagnosis of Alzheimer's Disease (AD) will be randomized to receive either S-equol or placebo first, and then cross over to receive the opposite intervention. The study, therefore, consists of two treatment periods with randomly assigned treatment order. Specifically, subjects are randomized to either: (1) S-equol for one month, then placebo for one month; or (2) placebo for one month, then S-equol for one month.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Alzheimer's Disease (AD)
* Have a study partner who has a close relationship with the participant and will attend study visits with the participant
* Do not possess an Alkylphenol ethoxylates 4 (APOE4) variant of the APOE gene
* Speak English as their primary language
* Have not had any medication changes within the past 30 days

Exclusion Criteria:

* Reside in a nursing home or dementia special care unit
* Have a potentially confounding, serious medical risk such as insulin-requiring diabetes, any history of cancer that required a chemotherapy or radiation therapy intervention within the past 5 years, or a recent cardiac event
* Have any clinically significant abnormal safety laboratory values at the SEAD2 screening visit
* Have any clinically significant abnormal findings on vital signs measurements, or on physical or neurological examination at the SEAD2 screening visit
* Use any type of systemic estrogen or testosterone replacement therapy
* Has participated in another clinical trial or received any investigational drug or investigational therapy within 30 days before the screening visit

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Swerdlow, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - Clinical and Translational Science Unit, Fairway, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- S-equol First, Then Placebo: This was a cross-over study. Each participant acted as their own control. The order of the interventions was randomized. Each participant spent one month in each intervention arm. In this group, participants initially received S-equol for one month, and at the conclusion of that arm they were switched to the placebo for one month. There was no washout period. The S-equol was provided as 50 mg capsules, which were taken twice daily.
- Placebo First, Then S-equol: This was a cross-over study. Each participant acted as their own control. The order of the interventions was randomized. Each participant spent one month in each intervention arm. In this group, participants initially received placebo for one month, and at the conclusion of that arm they were switched to S-equol for one month. There was no washout period. The S-equol was provided as 50 mg capsules, which were taken twice daily.
Period: Overall Study
Arm/Group | S-equol First, Then Placebo | Placebo First, Then S-equol
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- S-equol First, Then Placebo: This group received S-equol for one month, and then crossed over to receive placebo for one month. There was no washout period.
- Placebo First, Then S-Equol: This group received placebo for one month, then crossed over to receive S-equol for one month. There was no washout period.
- Total: Total of all reporting groups
Arm/Group | S-equol First, Then Placebo | Placebo First, Then S-Equol | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.7 (7.2) | 71.7 (8.4) | 74.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 11 | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 18 | 20 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cytochrome Oxidase/Citrate Synthase (COX/CS) Activity
Description: Cytochrome oxidase (COX) was measured in platelet mitochondria as a pseudo-first order rate constant (sec-1/mg protein), which was determined as a Vmax, spectrophotometrically, by tracking the change in absorbance as reduced cytochrome c is oxidized to oxidized cytochrome C. Citrate synthase (CS) is a soluble mitochondrial matrix enzyme whose activity was determined spectrophotometrically as a Vmax (micromoles/mg protein). Reporting the COX activity as a ratio to CS activity takes mitochondrial mass into account, and normalizes the COX activity per the amount of mitochondria present in the assay sample, with units 1/(seconds multiplied by micromoles).
Time Frame: Column 1 is the value after completing S-equol minus the value after completing placebo. For S-equol then placebo, this is the Visit 3 minus the Visit 4 COX/CS value. For placebo then S-equol, this is the Visit 4 minus the Visit 3 COX/CS value.
Population: Due to the pandemic, 1 participant in the Placebo, Then S-equol group did not complete the analysis. This subject was excluded from this primary analysis, and all secondary analyses except for the safety analysis. As the order of the intervention does not matter, all 39 participants who contributed COX/CS data to the final analysis are included. The mean (SD) value reflects the mean of values obtained when the COX/CS value while on placebo was subtracted from the COX/CS score while on S-equol.
Measure: Mean (Standard Deviation); unit: 1/(seconds multiplied by micromoles)
Groups:
- Difference (on S-equol Minus on Placebo): Value after completion of S-equol minus value after completion of placebo. For S-equol then placebo, this is the Visit 3 minus the Visit 4 COX/CS value. For placebo then S-equol, this is the Visit 4 minus the Visit 3 COX/CS value.
- S-equol: This is the average COX/CS measured after S-equol (at month 3 for those on S-equol then Placebo, at month 4 for those on Placebo then S-equol)
- Placebo: This is the average COX/CS measured after Placebo (at month 3 for those on Placebo then S-equol, at month 4 for those on S-equol then Placebo)
Arm/Group | Difference (on S-equol Minus on Placebo) | S-equol | Placebo
Number analyzed (Participants) | 39 | 39 | 39
1/(seconds multiplied by micromoles) | -0.0000049 (0.000024) | 0.0000195 (0.0000081) | 0.0000245 (0.0000258)
Statistical Analysis 1: Comparison: Difference (on S-equol Minus on Placebo); As the order of the intervention does not matter, all 39 participants who contributed data to the final analysis are included together; Test type: Other — We performed a paired T-test analysis to ascertain whether the COX/CS activity while on S-equol was comparable or different than the COX/CS while on placebo. For each participant, the COX/CS value while on S-equol was subtracted from their COX/CS value while on placebo; p > 0.05, Paired T-test

2. Secondary Outcome: Pattern of COX Activity Changes While on the Active Treatment Versus Placebo Arms of This Crossover Study.
Description: Participants are defined as responders or non-responders depending on the slope of COX/CS activity change. Those in the "Responder" group have a greater slope of COX/CS activity change going from off- to on-S-equol as compared to going from on- to off-S-equol.
Time Frame: Visits 2, 3, 4
Population: Only the 20 participants who had baseline then S-equol then placebo values contributed to this analysis.
Measure: Number; unit: participants
Groups:
- S-equol Then Placebo Subjects Only: Only subjects that received S-equol then placebo were used for this analysis. Those that received placebo then S-equol were excluded from this analysis.
Arm/Group | S-equol Then Placebo Subjects Only
Number analyzed (Participants) | 20
participants | 7

3. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: Scale range: 0-30. A higher score indicates better global cognitive performance.
Time Frame: Score after completion of S-equol minus score after completion of placebo. For S-equol then placebo, this is the Visit 3 minus the Visit 4 MoCA score. For placebo then S-equol, this is the Visit 4 minus the Visit 3 MoCA score.
Population: The one subject missing the COX/CS difference score was excluded from this analysis. The key measure is the difference score. Participants unable to contribute both S-equol and placebo scores were not included in the difference score analysis, but do contribute to the S-equol or placebo scores as available.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Difference (on S-equol Minus on Placebo): This is the average within subject MoCA measure after S-equol minus after Placebo (at month 3 minus at month 4 for those on S-eqol then Placebo, at month 4 minus at month 3 for those on Placebo then S-equol)
- S-equol: This is the average MoCA measured after S-equol (at month 3 for those on S-equol then Placebo, at month 4 for those on Placebo then S-equol)
- Placebo: This is the average MoCA measured after Placebo (at month 3 for those on Placebo then S-equol, at month 4 for those on S-equol then Placebo)
Arm/Group | Difference (on S-equol Minus on Placebo) | S-equol | Placebo
Number analyzed (Participants) | 35 | 35 | 36
score on a scale | 0.2 (2.4) | 12.3 (6.3) | 12.0 (6.1)

4. Secondary Outcome: Alzheimer's Disease Assessment Scale-Cognitive Portion (ADASCog-11)
Description: Scale range: 0-70. A lower score indicates better global cognitive performance.
Time Frame: Score after completion of S-equol minus score after completion of placebo. For S-equol then placebo, this is the Visit 3 minus the Visit 4 ADASCog score. For placebo then S-equol, this is the Visit 4 minus the Visit 3 ADASCog score.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Difference (on S-equol Minus on Placebo): This is the average within subject ADAS-Cog measure after S-equol minus after Placebo (at month 3 minus at month 4 for those on S-equol then Placebo, at month 4 minus at month 3 for those on Placebo then S-equol)
- S-equol: This is the average ADAS-Cog measured after S-equol (at month 3 for those on S-equol then Placebo, at month 4 for those on Placebo then S-equol)
- Placebo: This is the average ADAS-Cog measured after placebo (at month 3 for those on placebo then S-equol then Placebo, at month 4 for those on S-equol then Placebo
Arm/Group | Difference (on S-equol Minus on Placebo) | S-equol | Placebo
Number analyzed (Participants) | 36 | 36 | 36
score on a scale | 1.1 (5.5) | 24.6 (11.3) | 23.5 (10.6)

5. Secondary Outcome: Logical Memory Test 1 (LMT1) - Immediate Recall
Description: Scale range: 0-25. A higher score indicates better memory function.
Time Frame: Score after completion of S-equol minus score after completion of placebo. For S-equol then placebo, this is the Visit 3 minus the Visit 4 LMT1 score. For placebo then S-equol, this is the Visit 4 minus the Visit 3 LMT1 score.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Difference (on S-equol Minus on Placebo): Score after completion of S-equol minus score after completion of placebo. For S-equol then placebo, this is the Visit 3 minus the Visit 4 LMT1 score. For placebo then S-equol, this is the Visit 4 minus the Visit 3 LMT1 score.
- S-equol: This is the average LMT1 score measured after S-equol (at month 3 for those on S-equol then Placebo, at month 4 for those on Placebo then S-equol)
- Placebo: This is the average ADAS-Cog LMT1 score measured after S-equol (at month 3 for those on Placebo then S-equol, at month 4 for those on S-equol then Placebo)
Arm/Group | Difference (on S-equol Minus on Placebo) | S-equol | Placebo
Number analyzed (Participants) | 36 | 36 | 36
score on a scale | 0.2 (2.9) | 4.1 (4.2) | 3.9 (3.3)

6. Secondary Outcome: Logical Memory Test 2 (LMT2) - Delayed Recall
Description: Scale range: 0-25. A higher score indicates better memory performance.
Time Frame: Score after completion of S-equol minus score after completion of placebo. For S-equol then placebo, this is the Visit 3 minus the Visit 4 LMT2 score. For placebo then S-equol, this is the Visit 4 minus the Visit 3 LMT2 score.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Difference (on S-equol Minus on Placebo): Score after completion of S-equol minus score after completion of placebo. For S-equol then placebo, this is the Visit 3 minus the Visit 4 LMT2 score. For placebo then S-equol, this is the Visit 4 minus the Visit 3 LMT2 score.
- S-equol: This is the average LMT2 measured after S-equol (at month 3 for those on S-equol then Placebo, at month 4 for those on Placebo then S-equol)
- Placebo: This is the average LMT2 measured after Placebo (at month 3 for those on Placebo then S-equol, at month 4 for those on S-equol S-equol then Placebo)
Arm/Group | Difference (on S-equol Minus on Placebo) | S-equol | Placebo
Number analyzed (Participants) | 36 | 36 | 36
score on a scale | 0.2 (2.0) | 1.9 (3.4) | 1.8 (2.7)

7. Secondary Outcome: Stroop Color Test Score
Description: Scale range: 0-unlimited. A higher score indicates better executive function.
Time Frame: Score after completion of S-equol minus score after completion of placebo. For S-equol then placebo, this is the Visit 3 minus the Visit 4 Stroop Color Test score. For placebo then S-equol, this is the Visit 4 minus the Visit 3 Stroop Color Test score.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Difference (on S-equol Minus on Placebo): Score after completion of S-equol minus score after completion of placebo. For S-equol then placebo, this is the Visit 3 minus the Visit 4 Stroop Color Test score. For placebo then S-equol, this is the Visit 4 minus the Visit 3 Stroop Color Test score.
- S-equol: This is the average Stroop Color Test score measured after S-equol (at month 3 for those on S-equol then Placebo, at month 4 for those on Placebo then S-equol)
- Placebo: This is the average Stroop Color Test score measured after S-equol (at month 3 for those on Placebo then S-equol, at month 4 for those on S-equol then Placebo)
Arm/Group | Difference (on S-equol Minus on Placebo) | S-equol | Placebo
Number analyzed (Participants) | 34 | 34 | 35
score on a scale | -0.1 (5.8) | 40.0 (20.9) | 39.3 (18.5)

8. Secondary Outcome: Stroop Word Test
Description: Scale range: 0-unlimited. A higher score indicates better executive function.
Time Frame: Score after completion of S-equol minus score after completion of placebo. For S-equol then placebo, this is the Visit 3 minus the Visit 4 Stroop Word Test score. For placebo then S-equol, this is the Visit 4 minus the Visit 3 Stroop Word Test score.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Difference (on S-equol Minus on Placebo): Score after completion of S-equol minus score after completion of placebo. For S-equol then placebo, this is the Visit 3 minus the Visit 4 Stroop Word score. For placebo then S-equol, this is the Visit 4 minus the Visit 3 Stroop Word score.
- S-equol: This is the average Stroop Word score measured after S-equol (at month 3 for those on S-equol then Placebo, at month 4 for those on Placebo then S-equol)
- Placebo: This is the average Stroop Word score measured after placebo (at month 3 for those on Placebo then S-equol, and at month 4 for those on S-equol then placebo)
Arm/Group | Difference (on S-equol Minus on Placebo) | S-equol | Placebo
Number analyzed (Participants) | 35 | 35 | 35
score on a scale | -0.1 (9.5) | 56.1 (23.1) | 56.3 (21.9)

9. Secondary Outcome: Stroop Interference Test
Description: Scale range: 0-unlimited. A higher score indicates better executive function.
Time Frame: Score after completing S-equol minus score after completing placebo. For S-equol then placebo, this is the Visit 3 minus the Visit 4 Stroop Interference score. For placebo then S-equol, this is the Visit 4 minus the Visit 3 Stroop Interference score.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Difference (on S-equol Minus on Placebo): Score after completion of S-equol minus score after completion of placebo. For S-equol then placebo, this is the Visit 3 minus the Visit 4 Stroop Interference score. For placebo then S-equol, this is the Visit 4 minus the Visit 3 Stroop Interference score.
- S-equol: This is the average Stroop Interference score measured after S-equol (at month 3 for those on S-equol then Placebo, at month 4 for those on Placebo then S-equol)
- Placebo: This is the average Stroop Interference score measured after Placebo (at month 3 for those on Placebo then S-equol, at month 4 for those on S-equol then Placebo)
Arm/Group | Difference (on S-equol Minus on Placebo) | S-equol | Placebo
Number analyzed (Participants) | 28 | 28 | 29
score on a scale | -1.2 (6.8) | 14.5 (7.4) | 15.3 (8.2)

10. Secondary Outcome: Number of Participants With Adverse Events
Description: List of adverse events as reported over the course of the study (safety labs, physical and neurological exams, vital signs, signs and symptoms).
Time Frame: 4 Months: From Visit 1 (Day 0) through Visit 1 (end of month 1, +/- 7 days), Visit 2 (end of month 2, +/- 7 days), Visit 3 (end of month 3, +/- 7days), and Post-Interventions Phone Call (end of month 4, +/- 7 days)
Population: All 40 enrolled participants contributed to the safety data
Measure: Number; unit: participants
Groups:
- Prior to Starting Drug or Placebo: This group applies to the Lead-in period, which includes the period 1 month (+/- 7 days) between the screening visit and starting the first intervention.
- While on S-equol: This group includes adverse events while on S-equol, regardless of treatment order. Some received S-equol then placebo, and some received placebo then S-equol. All subjects contributed to each group; 20 who started on S-equol and crossed over to placebo, and 20 who started on placebo and crossed over to S-equol. 40 represents the sum of both these arms, as all received S-equol.
- While on Placebo: This group includes adverse events while on placebo, regardless of treatment order. Some received S-equol then placebo, and some received placebo then S-equol. All subjects contributed to each group; 20 who started on S-equol and crossed over to placebo, and 20 who started on placebo and crossed over to S-equol. 40 represents the sum of both these arms, as all received placebo.
- After Completing Both Drug and Placebo: This applies to the post-interventions observation period, which took place 1 month (+/- 7 days) after completing the second intervention arm.
Arm/Group | Prior to Starting Drug or Placebo | While on S-equol | While on Placebo | After Completing Both Drug and Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40
participants | 1 | 8 | 8 | 4

ADVERSE EVENTS:
Time Frame: 4 months: From Visit 1 (Day 0) through Visit 1 (end of month 1, +/- 7 days), Visit 2 (end of month 2, +/- 7 days), Visit 3 (end of month 3, +/- 7days), and Post-Interventions Phone Call (end of month 4, +/- 7 days)
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- Prior to Starting Drug or Placebo: This includes all 40 participants, prior to the initiation of any treatment (S-equol or placebo).
- While on S-equol: This includes all 40 participants while receiving S-equol 50mg twice daily for one month.
- While on Placebo: This includes all 40 participants while receiving placebo twice daily for one month.
- After Completing Both Drug and Placebo: This includes all 40 participants following completion of their courses of both S-equol and placebo, regardless of treatment order.
Arm/Group | Prior to Starting Drug or Placebo | While on S-equol | While on Placebo | After Completing Both Drug and Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 1/40 | 8/40 | 8/40 | 4/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Prior to Starting Drug or Placebo (N=40) | While on S-equol (N=40) | While on Placebo (N=40) | After Completing Both Drug and Placebo (N=40)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal Acid Reflux (Gastrointestinal disorders) | 0/0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fecal Impaction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Pressure Change (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vasovagal Event (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bruise (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth Extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retina Procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased Urinary Frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney Stone (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Viral Respiratory Infection/Cold (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gum Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT03101085/Prot_SAP_000.pdf